CLINICAL TRIAL: NCT06936904
Title: Impact of Different Injection Rate on Local Anaesthetic Spread of Ultrasound-guided Erector Spinae Plane Block
Brief Title: Different Injection Speed on Local Anaesthetic Spread of ESPB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Tao Shan, Attending physician, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20250327-16
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Erector Spinae Plane Block

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Other): A total of 30 ml of the local anesthetic solution (0.375% ropivacaine, comprising 15 ml ropivacaine and 15 ml iodinated contrast) is injected. In the Group C, the injection is administered within 180 seconds.
  Interventions: Procedure: injection speed
- Group S (Experimental): A total of 30 ml of the local anesthetic solution (0.375% ropivacaine, comprising 15 ml ropivacaine and 15 ml iodinated contrast) is injected. In the Group S, the injection is administered within 30 seconds.
  Interventions: Procedure: injection speed

INTERVENTIONS:
Procedure: injection speed — Patients undergoing CT-guided lung nodule localization were selected for the study, and ultrasound-guided erector spinae plane block was performed before surgery with different injection speed.

SUMMARY:
The aim of this clinical trial is to investigate the effect of different injection speeds on the spread of local anesthetic during ultrasound-guided erector spinae plane block (ESPB) in patients undergoing CT-guided lung nodule localization. The primary question addressed is whether a high injection speed (30 ml delivered within 30 seconds) produces a different local anesthetic distribution compared with a lower injection speed (30 ml delivered within 180 seconds).

DETAILED DESCRIPTION:
Senventy-four patients were selected to undergo CT guided puncture localization of lung nodules under local anesthesia, and the patients were divided into groups using a computer-generated random number in a ratio of 1:1. To ensure objectivity, a nurse who was not involved in the study prepared a sealed opaque envelope containing grouping information. Patients were randomly divided into two groups: control group (group C, 37 patients), and experimental group (group S, 37 patients). All patients underwent ultrasound guided ESPB before CT-guided nodule localization. Ultrasound guided ESPB method: Using a high-frequency linear probe (5-13 MHz, Sonosite, USA), the probe is placed parallel to the spine on the surface of the transverse process tip of the seventh thoracic vertebrae. Under ultrasound, the transverse process and spinal muscles are clearly exposed. Then, a long beveled needle is used, and inserted from the cephalad to caudal with in-plane technique. After the needle tip reaches between the transverse process and erector spinae muscles, 2ml saline is injected using water separation technique to confirm the position of the needle tip, then injecting 30ml local anesthetic solution (0.75% ropivacaine 15ml+iohexol 15ml). In the control group, the injection is administered at a rate of 30 ml within 180 seconds. In the experimental group, the injection is delivered at a faster rate of 30 ml withinr 30 seconds. After 30 minutes of block completion, CT scan and puncture localization were performed, following with 3D reconstruction. The primary outcome was mixture spread to the paravertebral space.The second outcomes were as follow: 1.spread to the intercostal space. 2. spread to the epidural space 3.spread to the neural foramina 4. cranio-caudal spread

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for CT-guided lung nodule localization under local anesthesia will be selected

1. aged 18-80 years
2. BMI 18-30 kg/m²
3. ASA classification I-III

Exclusion Criteria:

1. Allergy to the study drug or to local anesthetics
2. History of opioid abuse
3. Previous infection at the ESPB or PVB puncture site
4. Peripheral neuropathy
5. Dysfunction of blood coagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Spread of local anesthetic into the paravertebral space | 30 minutes after completion of the ESPB block
  Observation of local anesthetic spread into the paravertebral space with CT by a researcher who was blinded to group allocation

SECONDARY OUTCOMES:
Diffusion of local anesthetic into intercostal space | 30 minutes after completion of the block
  The Incidence and thoracic level of local anesthetics to intercostal space was observed with CT by a researcher who was blinded to group allocation.
Diffusion of local anesthetic into the epidural space | 30 minutes after completion of the block
  Incidence and segment of local anesthetic spread into the epidural was assessed by a researcher who was blinded to group allocationTime Frame: 30 minute after completion of the block
Diffusion of local anesthetic into the neural foramina | 30 minutes after completion of the block
  Incidence and segment of local anesthetic spread into the neural foramina was assessed by a researcher who was blinded to group allocationTime Frame: 30 minute after completion of the block
Cephalocaudal spread of local anesthetic | 30 minutes after completion of the block
  Observation of local anesthetic spread cephalocaudally
Loss to Cold Sensation of Skin | 30 minutes after block
  The sensation to cold was assessed with ice. The area includes the anterior chest wall (midclavicular line), lateral chest wall (posterior axillary line), and posterior chest wall (paraspinal zone) by a researcher who was blinded to group allocation.
NRS (Numeric Rating Scales) Score | 1 hour after CT-guided nodule localization
  Numerical Rating Scale (NRS): This scale is composed of 11 numbers from 0 to 10, with higher numbers indicating greater pain intensity.Patients are required to select a number from 0 to 10 that best represents their current pain intensity based on patients' experience.
Hemodynamic profile | Heart rate changes before blockade, 5minute after blockade, 10 minute after blockade, 20minute after blockade, 30minute after blockade
  Hemodynamic changes(Heart rate ) during blockade procedure
Hemodynamic profile | Mean arterial pressure changes before blockade, 5minute after blockade, 10 minute after blockade, 20minute after blockade, 30minute after blockade
  Hemodynamic changes(Mean arterial pressure ) during blockade procedure

CONTACTS AND LOCATIONS:
Overall Officials: Tao Shan, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No